CLINICAL TRIAL: NCT05108779
Title: Phase Ia Clinical Study of Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of QLF32004 for Injection Monotherapy in Patients With Advanced Malignant Tumors
Brief Title: QLF32004 Injection for the Treatment of Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLF32004-101
Record Dates: First submitted 2021-10-22; First posted 2021-11-05 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-08

CONDITIONS: Advanced Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLF32004 (Experimental)
  Interventions: Drug: QLF32004

INTERVENTIONS:
Drug: QLF32004 — In the phase, five dose groups were proposed.The frequency of administration was once a week, and the treatment cycle was 3 weeks.

SUMMARY:
To determine the safety, tolerability, and recommended dose (RP2D) of QLF32004 in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old .
2. Patients with advanced malignant solid tumors confirmed histologically or cytologically have failed standard therapy, or have no standard therapy, or are not eligible for standard therapy at this stage.
3. (dose escalation phase) At least one assessable tumor focus according to RECIST 1.1;(PK expansion phase) According to RECIST 1.1, there is at least one measurable tumor lesion (a tumor lesion located in the area of previous radiotherapy or other local regional treatment site is generally not considered measurable unless the lesion shows definite progression or persists after 3 months of radiotherapy).
4. ECOG score 0-1.
5. Life expectancy ≥ 12 weeks.
6. Adequate organ function prior to the first use of the investigational drug (no use of any blood components, cell growth factor, colony stimulating factor (G-CSF), rhTPO, etc., or hepatoprotective therapy is permitted within 14 days prior to laboratory examination);
7. Eligible fertile patients (male and female) must agree to use a reliable contraceptive method (hormonal or barrier methods or abstinence, etc.) with their partner during the trial and for 6 months after the last medication;Women of reproductive age must have a negative blood pregnancy test within 7 days of their first use of the study drug;
8. Subjects shall give informed consent to this study before the test and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Known allergy to the study drug or any excipients thereof; Or had a grade ≥3 allergic reaction to protein drugs in the past.
2. Had received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks prior to the first use of the study drug.
3. Received any other investigational drug or treatment that is not on the market within 4 weeks prior to the first use of the investigational drug.
4. Use of live attenuated vaccine within 4 weeks prior to initial use of the study drug.
5. Received systemic glucocorticoid or other immunosuppressant treatment within 14 days prior to initial use of the study drug.
6. Use of immunomodulatory drugs, including but not limited to thymosin.
7. Had major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to initial use of the study drug, or required elective surgery during the study period.
8. Patients with cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms were judged by the investigator to be unsuitable for inclusion;
9. Patients with uncontrollable exudation (thorax, pericardium, abdominal cavity);
10. Have received immunotherapy and present with grade ≥ 3 irAE or grade ≥2 immune-associated myocarditis;
11. Adverse reactions of previous antitumor therapy have not recovered to CTCAE 5.0 rating ≤1 (except toxicity without safety risk, such as hair loss, peripheral neurotoxicity of grade 2, hypothyroidism stabilized by hormone replacement therapy, etc.);
12. Presence or history of any active autoimmune disease;Subjects with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, hair loss, type I diabetes, or asthma that has been completely resolved in childhood and does not require any intervention as adults may be included;Asthma patients requiring medical intervention with bronchodilators were excluded;
13. Patients with previous or current interstitial lung disease;
14. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); Active hepatitis B, active hepatitis C;

16. Have a history of serious cardiovascular and cerebrovascular diseases; 17. Have active infection and currently require intravenous anti-infection therapy; 18. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 19. The patient is known to have a history of psychotropic drug abuse, alcoholism or drug abuse;A clear past history of neurological or psychiatric disorders, including epilepsy or dementia; 20. Patients with other serious physical or mental disorders or abnormal laboratory tests that may increase the risk of study participation or interfere with study results, and who are considered unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 21 days
Maximum Tolerated Dose (MTD) | 21 days
Recommended Phase 2 Dose (RP2D) | 12 month

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | 21 days
Maximum Observed Plasma Concentration (Cmax) | 21 days
Serious Adverse Event (SAE) | 12 month
Area Under The Curve (AUC) | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China